CLINICAL TRIAL: NCT02177032
Title: Phase 3, Randomized, Stratified, Open Label, Multicenter, Controlled Clinical Study to Evaluate Safety and Immunogenicity of a Rabies Vaccine Administered, With and Without Human Rabies Immunoglobulin, Using the New "4-sites, 1-week" Intradermal Regimen for Postexposure Prophylaxis Compared to the Currently Recommended "2-sites, TRC" Intradermal Regimen in Children and Adults Subjects.
Brief Title: Safety and Immunogenicity of Two Intradermal Rabies Vaccine Regimens Administered With and Without Human Rabies Immunoglobulin in Subjects ≥ 1 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V49_30; 2013-CT0191 (Registry Identifier: registry.healthresearch.ph)
Record Dates: First submitted 2014-06-24; First posted 2014-06-27 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-02

CONDITIONS: Rabies Infection
Keywords: Rabies vaccines; intradermal; human rabies immunoglobulins
MeSH Terms: interventions — Rabies Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 4-sites, 1-week without HRIG (Experimental): PCEC rabies vaccine, administered ID according to the "4-sites, 1-week" regimen
  Interventions: Biological: Rabies vaccine
- 4-sites, 1-week with HRIG (Experimental): PCEC rabies vaccine, administered ID to adults, according to the "4-sites, 1-week" regimen plus HRIG
  Interventions: Biological: Rabies vaccines + Rabies immunoglobulins
- 2-sites, TRC without HRIG (Active Comparator): PCEC rabies vaccine, administered ID according to the "2-sites, TRC" regimen
  Interventions: Biological: Rabies vaccine
- 2-sites, TRC with HRIG (Active Comparator): PCEC rabies vaccine, administered ID to adults , according to the "2-sites, TRC" regimen plus HRIG
  Interventions: Biological: Rabies vaccines + Rabies immunoglobulins

INTERVENTIONS:
Biological: Rabies vaccine — 12 doses of the PCEC rabies vaccine, administered ID (0.1mL for each injection) according to the "4-sites, 1-week" regimen (i.e. 4 doses of vaccine; in both deltoids and anterolateral thigh areas, administered on days 1, 4, and 8).
  Arms: 4-sites, 1-week without HRIG
Biological: Rabies vaccines + Rabies immunoglobulins — 12 doses of the PCEC rabies vaccine, administered ID (0.1mL for each injection) to adults only, according to the "4-sites, 1-week" regimen (i.e. 4 doses of vaccine; in both deltoids and anterolateral thigh areas, administered on days 1, 4, and 8). HRIG will be administered on day 1 (before the first dose of the vaccine) in a dose of 20 IU/kg body weight intramuscularly into the gluteal muscle.
  Arms: 4-sites, 1-week with HRIG
Biological: Rabies vaccine — 8 doses of the PCEC rabies vaccine, administered ID (0.1ml for each injection) according to the "2-sites, TRC", updated Thai Red Cross regimen (i.e. 2 doses of vaccine; in both deltoids, administered on days 1, 4, 8, and 29).
  Arms: 2-sites, TRC without HRIG
Biological: Rabies vaccines + Rabies immunoglobulins — 8 doses of the PCEC rabies vaccine, administered ID (0.1ml for each injection) to adults only, according to the "2-sites, TRC", updated Thai Red Cross regimen (i.e. 2 doses of vaccine; in both deltoids, administered on days 1, 4, 8, and 29). HRIG will be administered on day 1 (before the first dose of the vaccine) in a dose of 20 IU/kg body weight intramuscularly into the gluteal muscle.
  Arms: 2-sites, TRC with HRIG

SUMMARY:
Demonstrate non-inferiority of the immune response between new versus the currently recommended intradermal regimens of rabies vaccine when administered with or without rabies immunoglobulins in healthy subjects ≥ 1 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females ≥ 1 years of age
2. Individuals/ individual's parents or legal guardians who have given written consent
3. Individuals in good health
4. Individuals who can comply with study procedures

Exclusion Criteria:

1. Behavioral or cognitive impairment or psychiatric disease.
2. Unable to comprehend and to follow all required study procedures for the whole period of the study.
3. History of illness or with an ongoing illness that may pose additional risk to the individual if he/she participates in the study.
4. Individuals ≥ 1 to ≤ 17 years of age, who have or ever had a malignancy.
5. Individuals ≥ 18 years of age, who have or who within the last 5 years, have had a malignancy (excluding nonmelanotic skin cancer) or lymphoproliferative disorder.
6. Known or suspected impairment of the immune system (including but not limited to HIV, autoimmune disorders, immunosuppressive therapy as applicable).
7. Female of childbearing potential who has not used any of the "acceptable contraceptive methods" for at least 2 months prior to study entry.
8. Female of childbearing potential, refusal to use an "acceptable birth control method" through day 50.
9. Female of childbearing potential, with a positive pregnancy test prior to enrollment.
10. Received blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation in the previous 12 weeks.
11. Allergic to any of the vaccine components.
12. Allergic to any of the human rabies immunoglobulin components.
13. Contraindication or precaution against rabies vaccination.
14. Contraindication or precaution against man rabies immunoglobulin administration.
15. Planning to receive anti-malaria medications (e.g. Mefloquine) 14 days prior to day 1 vaccination through day 50.
16. Participating in any clinical trial with another investigational product 30 days prior to first study visit or intent to participate in another clinical study at any time during the conduct of this study.
17. Received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this study or who are planning to receive any vaccine within 28 days from the study vaccines.
18. Body temperature ≥ 38.0°C (≥ 100.4°F) within 3 days of intended study vaccination.
19. Received rabies vaccines or rabies immunoglobulin or have been exposed to rabies.
20. Part of the study personnel or immediate family members of study personnel conducting this study.
21. Current or history of drug or alcohol abuse within the past 2 years.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 885 (Actual)
Dates: Start 2014-06; Primary Completion 2014-10 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (6):
- Philippines (4):
  - 4, De La Salle Health Sciences Institute, Cavite
  - 1, Research Institute for Tropical Medicine, City of Muntinlupa
  - 2, Asian Hospital and Medical Center, City of Muntinlupa
  - 3, Research Institute for Tropical Medicine, City of Muntinlupa
- Thailand (2):
  - 11, Infectious Diseases Unit, Department of Pediatrics, Phramongkutklao hospital, Bangkok, Bangkok
  - 12, Department of Tropical Pediatrics, Faculty of Tropical Medicine, Mahidol University, Bangkok, Bangkok

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- 4-sites, 1-week WITHOUT HRIG: 12 doses of the PCEC rabies vaccine, administered ID (0.1mL for each injection) according to the "4-sites, 1-week" regimen
- 4-sites, 1-week WITH HRIG: 12 doses of the PCEC rabies vaccine, administered ID (0.1mL for each injection) to adults only, according to the "4-sites, 1-week" regimen HRIG administered on day 1 (before the first dose of the vaccine) in a dose of 20 IU/kg body weight intramuscularly
- 2-sites, TRC WITHOUT HRIG: 8 doses of the PCEC rabies vaccine, administered ID (0.1ml for each injection) according to the "2-sites, TRC", updated Thai Red Cross regimen
- 2-sites, TRC WITH HRIG: 8 doses of the PCEC rabies vaccine, administered ID (0.1ml for each injection) to adults only, according to the "2-sites, TRC", updated Thai Red Cross regimen. HRIG administered on day 1 (before the first dose of the vaccine) in a dose of 20 IU/kg body weight intramuscularly
Period: Overall Study
Arm/Group | 4-sites, 1-week WITHOUT HRIG | 4-sites, 1-week WITH HRIG | 2-sites, TRC WITHOUT HRIG | 2-sites, TRC WITH HRIG
Started | 355 | 88 | 354 | 88
Completed | 350 | 86 | 351 | 88
Not Completed | 5 | 2 | 3 | 0
Not completed — ADMINISTRATIVE REASON | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0
Not completed — OTHER | 2 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- 4-sites, 1-week WITH HRIG: 12 doses of the PCEC rabies vaccine, administered ID (0.1mL for each injection) to adults only, according to the "4-sites, 1-week" regimen HRIG administered on day 1 (before the first dose of the vaccine) in a dose of 20 IU/kg body weight
- Total: Total of all reporting groups
Arm/Group | 4-sites, 1-week WITHOUT HRIG | 4-sites, 1-week WITH HRIG | 2-sites, TRC WITHOUT HRIG | 2-sites, TRC WITH HRIG | Total
Number analyzed (Participants) | 355 | 88 | 354 | 88 | 885
Age, Continuous [Mean (Standard Deviation); unit: year] | 20.0 (15.0) | 32.7 (10.8) | 20.6 (15.1) | 34.4 (11.2) | 22.9 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  FEMALE | 202 | 44 | 179 | 51 | 476
  MALE | 153 | 44 | 175 | 37 | 409

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With RVNA Titer >= 0.5 and Vaccine Group Differences ("4-sites, 1-week" to That of "2-sites, TRC" ID PEP Regimen of the PCEC Rabies Vaccine With or Without HRIG Administration)
Description: Vaccine group differences are calculated assuming a binomial distribution and the associated confidence interval for the differences in percentage was based on M-N method.
  Non-inferiority of the immune response of the new "4-sites, 1-week" ID PEP regimen of the PCEC vaccine, with or without HRIG administration, to that of the currently recommended "2-sites, TRC" ID PEP regimen of the PCEC rabies vaccine with or without HRIG administration, as measured by the percentage of subjects with RVNA titer ≥ 0.5 IU/ml at day 50 in the whole study population.
Time Frame: Study day 50 (D50)
Population: Per Protocol Set (PPS): all subjects who correctly receive the vaccine doses, provided immunogenicity data at the relevant time points and were not excluded due to reasons defined prior to the analysis.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Groups:
- TOTAL 4-sites, 1-week: 12 doses of the PCEC rabies vaccine, administered ID (0.1mL for each injection) to adults only, according to the "4-sites, 1-week" regimen with and without HRIG administered on day 1
- TOTAL 2-sites, TRC: 8 doses of the PCEC rabies vaccine, administered ID (0.1ml for each injection) to adults only, according to the "2-sites, TRC", updated Thai Red Cross regimen, with or without HRIG administered on day 1
Arm/Group | TOTAL 4-sites, 1-week | TOTAL 2-sites, TRC
Number analyzed (Participants) | 357 | 350
Percentages of Subjects | 99 [98 to 100] | 100 [99 to 100]
Statistical Analysis 1: Comparison: TOTAL 4-sites, 1-week vs TOTAL 2-sites, TRC; Test type: Non-Inferiority or Equivalence — The non-inferiority in immune response of the "4-sites, 1-week" (4-4-4-0-0) ID PEP regimen compared to the currently recommended "2-sites TRC" (2-2-2-0-2) ID PEP regimen, with or without HRIG, will be established If the lower bound of the two sided 95% confidence interval around the differences of the percentage of subject with RVNA titer ≥ 0.5 IU/ml at day 50 is > -0.05 (non-inferiority margin); Fisher Exact; Protection Rate Differences = -1, 95% CI 2-sided [-2.4 to 0]

2. Secondary Outcome: Geometric Mean Rabies Virus Neutralizing Antibody (RVNA) Concentration and Between-group (2 ID Rabies Vaccine Regimens (4-sites, 1-week and 2-sites, TRC) With or Without HRIG) Ratio of GMCs
Description: Immunogenicity was assessed in terms of Geometric Mean Rabies Virus Neutralizing Antibody (RVNA) Concentration in Children and Adult Subjects, ≥ 1 Years of Age at day 50 The GMCs, GMRs (i.e., within group ratio) and associated two sided 95% confidence intervals for each group were computed by exponentiating (base 10) of the least square means of the logarithmically transformed (base 10) concentration (and their differences) and the 95% CIs obtained from an Analysis of variance (ANOVA) with vaccine regimen, age strata and center as factors.
  Non-inferiority of the immune response between the 2 ID rabies vaccine regimens (4-sites, 1-week and 2-sites, TRC) with or without HRIG administration as measured by RVNA GMCs at day 50 in the whole study population.
Time Frame: Study Day 50
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Groups:
- TOTAL 4-sites, 1-week: 12 doses of the PCEC rabies vaccine, administered ID (0.1mL for each injection) according to the "4-sites, 1-week" regimen (i.e. 4 doses of vaccine; in both deltoids and anterolateral thigh areas, administered on days 1, 4, and 8) with or without HRIG administration on day 1
Arm/Group | TOTAL 4-sites, 1-week | TOTAL 2-sites, TRC
Number analyzed (Participants) | 357 | 350
IU/mL | 4.58 [4.15 to 5.06] | 10 [9.29 to 11]
Statistical Analysis 1: Comparison: TOTAL 4-sites, 1-week vs TOTAL 2-sites, TRC; Test type: Non-Inferiority or Equivalence — The investigational regimen 4-sites, 1-week" ID PEP will be declared as non-inferior to currently recommended "2-sites TRC" ID PEP regimen if the lower bound of the two sided 95% confidence interval around of the observed GMC ratio is greater than 0.667; ANOVA; Vaccine Group Ratios = 0.46, 95% CI 2-sided [0.37 to 0.58]

3. Secondary Outcome: Geometric Mean Rabies Virus Neutralizing Antibody Concentration at Days 8, 15, 91, 181 and 366 & Between-group (2 ID Rabies Vaccine Regimens (4-sites,1-week & 2-sites, TRC) With or Without HRIG) Ratio of GMCs in Children & Adult Subjects,≥ 1 Years of Age
Description: Immunogenicity was assessed in terms of the Geometric Mean Rabies Virus Neutralizing Antibody (RVNA) Concentration at Days 8, 15, 91, 181 and 366 in Children and Adult Subjects, ≥ 1 Years of Age The GMCs, GMRs (i.e., within group ratio) and associated two sided 95% confidence intervals for each group were computed by exponentiating (base 10) of the least square means of the logarithmically transformed (base 10) concentration (and their differences) and the 95% CIs obtained from an Analysis of variance (ANOVA) with vaccine regimen, age strata and center as factors.
  Non-inferiority of the immune response between the 2 ID rabies vaccine regimens (4-sites, 1-week and 2-sites, TRC) with or without HRIG administration as measured by RVNA GMCs at day 50 in the whole study population.
Time Frame: At Days 8, 15, 91, 181 and 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | TOTAL 4-sites, 1-week | TOTAL 2-sites, TRC
Number analyzed (Participants) | 363 | 362
IU/mL
  Day 8 (N= 363, 362) | 0.23 [0.21 to 0.25] | 0.14 [0.13 to 0.15]
  Day 15 (N= 357, 361) | 18 [17 to 20] | 12 [10 to 13]
  Day 91 (N= 358, 362) | 2.32 [2.09 to 2.56] | 3.68 [3.32 to 4.07]
  Day 181 (N= 357, 360) | 1.59 [1.41 to 1.78] | 1.44 [1.28 to 1.62]
  Day 366 (N= 356, 352) | 1.59 [1.41 to 1.79] | 1.14 [1.01 to 1.28]
Statistical Analysis 1: Comparison: TOTAL 4-sites, 1-week vs TOTAL 2-sites, TRC; Test type: Non-Inferiority or Equivalence — The investigational regimen 4-sites, 1-week" ID PEP will be declared as non-inferior to currently recommended "2-sites TRC" ID PEP regimen if the lower bound of the two sided 95% confidence interval around of the observed GMC ratio is greater than 0.667 (Day 8); ANOVA; Vaccine Group Ratios = 1.04, 95% CI 2-sided [0.84 to 1.29]
Statistical Analysis 2: Comparison: TOTAL 4-sites, 1-week vs TOTAL 2-sites, TRC; Test type: Non-Inferiority or Equivalence — The investigational regimen 4-sites, 1-week" ID PEP will be declared as non-inferior to currently recommended "2-sites TRC" ID PEP regimen if the lower bound of the two sided 95% confidence interval around of the observed GMC ratio is greater than 0.667 (Day 15); ANOVA; Vaccine Group Ratios = 1.68, 95% CI 2-sided [1.35 to 2.1]
Statistical Analysis 3: Comparison: TOTAL 4-sites, 1-week vs TOTAL 2-sites, TRC; Test type: Non-Inferiority or Equivalence — The investigational regimen 4-sites, 1-week" ID PEP will be declared as non-inferior to currently recommended "2-sites TRC" ID PEP regimen if the lower bound of the two sided 95% confidence interval around of the observed GMC ratio is greater than 0.667 (Day 91); ANOVA; Vaccine Group Ratios = 0.68, 95% CI 2-sided [0.54 to 0.85]
Statistical Analysis 4: Comparison: TOTAL 4-sites, 1-week vs TOTAL 2-sites, TRC; Test type: Non-Inferiority or Equivalence — The investigational regimen 4-sites, 1-week" ID PEP will be declared as non-inferior to currently recommended "2-sites TRC" ID PEP regimen if the lower bound of the two sided 95% confidence interval around of the observed GMC ratio is greater than 0.667 (Day 181); ANOVA; Vaccine Group Ratios = 1.22, 95% CI 2-sided [0.94 to 1.59]
Statistical Analysis 5: Comparison: TOTAL 4-sites, 1-week vs TOTAL 2-sites, TRC; Test type: Non-Inferiority or Equivalence — The investigational regimen 4-sites, 1-week" ID PEP will be declared as non-inferior to currently recommended "2-sites TRC" ID PEP regimen if the lower bound of the two sided 95% confidence interval around of the observed GMC ratio is greater than 0.667 (Day 366); ANOVA; Vaccine Group Ratios = 1.67, 95% CI 2-sided [1.27 to 2.19]

4. Secondary Outcome: Percentages of Subjects With Anti-RVNA Titer ≥0.5 IU/mL at Days 8, 15, 91, 181 and 366 in Children and Adult Subjects and Vaccine Group Differences (2 ID Rabies Vaccine Regimens (4-sites, 1-week and 2-sites, TRC), With or Without HRIG), ≥ 1 Years of Age
Description: Vaccine group differences are calculated assuming a binomial distribution and the associated confidence interval for the differences in percentage was based on M-N method.
  RVNA percentage of subjects with RVNA titer ≥ 0.5 IU/mL at study days 8, 15, 91, 181, and 366 following administration of the 2 ID rabies vaccine regimens (4-sites, 1-week and 2-sites, TRC), with or without HRIG, in the whole study population.
Time Frame: At Days 8, 15, 91, 181 and 366
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | TOTAL 4-sites, 1-week | TOTAL 2-sites, TRC
Number analyzed (Participants) | 363 | 362
Percentages of Subjects
  Day 8 (N= 363, 362) | 18 [15 to 23] | 10 [7 to 13]
  Day 15 (N= 357, 361) | 100 [99 to 100] | 100 [98 to 100]
  Day 91 (N= 358, 362) | 96 [94 to 98] | 99 [98 to 100]
  Day 181 (N= 357, 360) | 93 [90 to 95] | 93 [90 to 96]
  Day 366 (N= 356, 352) | 90 [86 to 93] | 83 [79 to 87]
Statistical Analysis 1: Comparison: TOTAL 4-sites, 1-week vs TOTAL 2-sites, TRC; Test type: Non-Inferiority or Equivalence — The non-inferiority in immune response of the "4-sites, 1-week" (4-4-4-0-0) ID PEP regimen compared to the currently recommended "2-sites TRC" (2-2-2-0-2) ID PEP regimen, with or without HRIG, will be established If the lower bound of the two sided 95% confidence interval around the differences of the percentage of subject with RVNA titer ≥ 0.5 IU/ml at Day 8 is > -0.05 (non-inferiority margin); Fisher Exact; Protection Rate Differences = 9, 95% CI 2-sided [3.8 to 13.9]
Statistical Analysis 2: Comparison: TOTAL 4-sites, 1-week vs TOTAL 2-sites, TRC; Test type: Non-Inferiority or Equivalence — The non-inferiority in immune response of the "4-sites, 1-week" (4-4-4-0-0) ID PEP regimen compared to the currently recommended "2-sites TRC" (2-2-2-0-2) ID PEP regimen, with or without HRIG, will be established If the lower bound of the two sided 95% confidence interval around the differences of the percentage of subject with RVNA titer ≥ 0.5 IU/ml at Day 15 is > -0.05 (non-inferiority margin); Fisher Exact; Protection Rate Differences = 0, 95% CI 2-sided [-1 to 1.6]
Statistical Analysis 3: Comparison: TOTAL 4-sites, 1-week vs TOTAL 2-sites, TRC; Test type: Non-Inferiority or Equivalence — The non-inferiority in immune response of the "4-sites, 1-week" (4-4-4-0-0) ID PEP regimen compared to the currently recommended "2-sites TRC" (2-2-2-0-2) ID PEP regimen, with or without HRIG, will be established If the lower bound of the two sided 95% confidence interval around the differences of the percentage of subject with RVNA titer ≥ 0.5 IU/ml at Day 91 is > -0.05 (non-inferiority margin); Fisher Exact; Protection Rate Differences = -3, 95% CI 2-sided [-6 to -1.4]
Statistical Analysis 4: Comparison: TOTAL 4-sites, 1-week vs TOTAL 2-sites, TRC; Test type: Non-Inferiority or Equivalence — The non-inferiority in immune response of the "4-sites, 1-week" (4-4-4-0-0) ID PEP regimen compared to the currently recommended "2-sites TRC" (2-2-2-0-2) ID PEP regimen, with or without HRIG, will be established If the lower bound of the two sided 95% confidence interval around the differences of the percentage of subject with RVNA titer ≥ 0.5 IU/ml at Day 181 is > -0.05 (non-inferiority margin); Fisher Exact; Protection Rate Differences = -1, 95% CI 2-sided [-4.5 to 3.2]
Statistical Analysis 5: Comparison: TOTAL 4-sites, 1-week vs TOTAL 2-sites, TRC; Test type: Non-Inferiority or Equivalence — The non-inferiority in immune response of the "4-sites, 1-week" (4-4-4-0-0) ID PEP regimen compared to the currently recommended "2-sites TRC" (2-2-2-0-2) ID PEP regimen, with or without HRIG, will be established If the lower bound of the two sided 95% confidence interval around the differences of the percentage of subject with RVNA titer ≥ 0.5 IU/ml at Day 366 is > -0.05 (non-inferiority margin); Fisher Exact; Protection Rate Differences = 6, 95% CI 2-sided [1.3 to 11.5]

5. Secondary Outcome: Geometric Mean Rabies Virus Neutralizing Antibody (RVNA) Concentration and Vaccine Group Differences in Adult Subjects, ≥ 18 Years of Age
Description: Immunogenicity was assessed in terms of the Geometric Mean Rabies Virus Neutralizing Antibody (RVNA) Concentration at Days 8, 15, 50,91, 181 and 366 in Adult Subjects, ≥ 18 Years of Age.
  RVNA GMCs with RVNA titer ≥ 0.5 IU/mL at days 8, 15, 50, 91, 181 and 366 and group differences (4-sites,1-week without HRIG versus 4-sites,1-week with HRIG; 4-sites,1-week with HRIG versus 2-sites,TRC with HRIG; 4-sites,1-week without HRIG versus 2-sites, TRC without HRIG)
Time Frame: At Days 8, 15, 50, 91, 181 and 366
Population: Per Protocol Set (PPS): all subjects who correctly receive the vaccine doses, provided immunogenicity data at the relevant time points and were not excluded due to reasons defined prior to the analysis. This outcome measure is applicable only for the 4-sites, 1-week with HRIG and 4-sites, 1-week without HRIG Groups.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Groups:
- 4-sites, 1-week WITH HRIG: 12 doses of the PCEC rabies vaccine, administered ID (0.1mL for each injection) to adults only, according to the "4-sites, 1-week" regimen with HRIG administered on day 1 (before the first dose of the vaccine) in a dose of 20 IU/kg body weight
Arm/Group | 4-sites, 1-week WITH HRIG | 4-sites, 1-week WITHOUT HRIG
Number analyzed (Participants) | 66 | 150
IU/mL
  Day 8 (N= 66, 150) | 0.21 [0.17 to 0.26] | 0.15 [0.13 to 0.17]
  Day 15 (N= 65, 146) | 13 [11 to 15] | 15 [13 to 17]
  Day 50 (N= 65, 146) | 1.97 [1.6 to 2.43] | 4.47 [3.9 to 5.13]
  Day 91 (N= 65, 149) | 1.01 [0.81 to 1.27] | 2.28 [1.96 to 2.65]
  Day 181 (N= 65, 146) | 0.88 [0.67 to 1.14] | 1.92 [1.61 to 2.29]
  Day 366 (N= 65, 145) | 0.68 [0.53 to 0.88] | 1.42 [1.19 to 1.69]
Statistical Analysis 1: Comparison: 4-sites, 1-week WITH HRIG vs 4-sites, 1-week WITHOUT HRIG; Test type: Non-Inferiority or Equivalence — The non-inferiority in immune response of the "4-sites, 1-week" (4-4-4-0-0) ID PEP regimen of the PCEC vaccine, with HRIG administration, compared to that of the new "4-sites, 1-week" (4-4-4-0-0) ID PEP regimen of the PCEC vaccine, without HRIG administration, in adult subjects will be established if the lower bound of the two sided 95% confidence interval around the differences of the percentage of subject with RVNA titer ≥ 0.5 IU/ml at Day 8 is > -0.05 (non-inferiority margin); Fisher Exact; Protection Rate Differences = -11, 95% CI 2-sided [-19.6 to -1]
Statistical Analysis 2: Comparison: 4-sites, 1-week WITH HRIG vs 4-sites, 1-week WITHOUT HRIG; Test type: Non-Inferiority or Equivalence — The non-inferiority in immune response of the "4-sites, 1-week" (4-4-4-0-0) ID PEP regimen of the PCEC vaccine, with HRIG administration, compared to that of the new "4-sites, 1-week" (4-4-4-0-0) ID PEP regimen of the PCEC vaccine, without HRIG administration, in adult subjects will be established if the lower bound of the two sided 95% confidence interval around the differences of the percentage of subject with RVNA titer ≥ 0.5 IU/ml at Day 15 is > -0.05 (non-inferiority margin); Fisher Exact; Protection Rate Differences = 0, 95% CI 2-sided [-5.6 to 2.6]
Statistical Analysis 3: Comparison: 4-sites, 1-week WITH HRIG vs 4-sites, 1-week WITHOUT HRIG; Test type: Non-Inferiority or Equivalence — The non-inferiority in immune response of the "4-sites, 1-week" (4-4-4-0-0) ID PEP regimen of the PCEC vaccine, with HRIG administration, compared to that of the new "4-sites, 1-week" (4-4-4-0-0) ID PEP regimen of the PCEC vaccine, without HRIG administration, in adult subjects will be established if the lower bound of the two sided 95% confidence interval around the differences of the percentage of subject with RVNA titer ≥ 0.5 IU/ml at Day 91 is > -0.05 (non-inferiority margin); Fisher Exact; Protection Rate Differences = -15, 95% CI 2-sided [-26 to -7.1]
Statistical Analysis 4: Comparison: 4-sites, 1-week WITH HRIG vs 4-sites, 1-week WITHOUT HRIG; Test type: Non-Inferiority or Equivalence — The non-inferiority in immune response of the "4-sites, 1-week" (4-4-4-0-0) ID PEP regimen of the PCEC vaccine, with HRIG administration, compared to that of the new "4-sites, 1-week" (4-4-4-0-0) ID PEP regimen of the PCEC vaccine, without HRIG administration, in adult subjects will be established if the lower bound of the two sided 95% confidence interval around the differences of the percentage of subject with RVNA titer ≥ 0.5 IU/ml at Day 181 is > -0.05 (non-inferiority margin); Fisher Exact; Protection Rate Differences = -17, 95% CI 2-sided [-29 to -7.1]
Statistical Analysis 5: Comparison: 4-sites, 1-week WITH HRIG vs 4-sites, 1-week WITHOUT HRIG; Test type: Non-Inferiority or Equivalence — The non-inferiority in immune response of the "4-sites, 1-week" (4-4-4-0-0) ID PEP regimen of the PCEC vaccine, with HRIG administration, compared to that of the new "4-sites, 1-week" (4-4-4-0-0) ID PEP regimen of the PCEC vaccine, without HRIG administration, in adult subjects will be established if the lower bound of the two sided 95% confidence interval around the differences of the percentage of subject with RVNA titer ≥ 0.5 IU/ml at Day 366 is > -0.05 (non-inferiority margin); Fisher Exact; Protection Rate Differences = -25, 95% CI 2-sided [-37.8 to -13.2]

6. Secondary Outcome: Percentages of Subjects With Anti-RVNA Titer ≥0.5 IU/mL in Adult Subjects, ≥ 18 Years of Age
Description: Immunogenicity was assessed in terms of the Percentages of Subjects With Anti-RVNA concentration ≥0.5 IU/mL at Days 8, 15, 50, 91, 181 and 366 in Adult Subjects, ≥ 18 Years of Age.
  Percentage of subjects with RVNA titer ≥ 0.5 IU/mL at days 8, 15, 50, 91, 181 and 366 and group differences (4-sites,1-week without HRIG versus 4-sites,1-week with HRIG; 4-sites,1-week with HRIG versus 2-sites,TRC with HRIG; 4-sites,1-week without HRIG versus 2-sites, TRC without HRIG)
Time Frame: At Days 8, 15,50, 91, 181 and 366
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 4-sites, 1-week WITH HRIG | 4-sites, 1-week WITHOUT HRIG
Number analyzed (Participants) | 66 | 151
Percentages of Subjects
  Day 1 (N= 66, 151) | 0 [0 to 5] | 0 [0 to 2]
  Day 8 (N= 66, 150) | 8 [3 to 17] | 19 [13 to 26]
  Day 15 (N= 65, 146) | 100 [94 to 100] | 100 [98 to 100]
  Day 50 (N= 65, 146) | 95 [87 to 99] | 100 [98 to 100]
  Day 91 (N= 65, 149) | 83 [72 to 91] | 98 [94 to 100]
  Day 181 (N= 65, 146) | 77 [65 to 86] | 94 [89 to 97]
  Day 366 (N= 65, 145) | 66 [53 to 77] | 91 [85 to 95]

7. Secondary Outcome: Geometric Mean Rabies Virus Neutralizing Antibody (RVNA) Concentration in Children and Adult Subjects, ≥ 1 Years of Age
Description: Immunogenicity was assessed in terms of the Geometric Mean Rabies Virus Neutralizing Antibody (RVNA) Concentration at Days 8, 15, 50, 91, 181 and 366 in Children and Adult Subjects, ≥ 1 Years of Age
Time Frame: At Days 8, 15, 50, 91, 181 and 366
Population: Per Protocol Set (PPS): all subjects who correctly receive the vaccine doses, provided immunogenicity data at the relevant time points and were not excluded due to reasons defined prior to the analysis. This outcome measure is applicable only for the 4-sites, 1-week without HRIG and 2-sites, TRC without HRIG Groups.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 4-sites, 1-week Without HRIG | 2-sites, TRC Without HRIG
Number analyzed (Participants) | 298 | 290
IU/mL
  Day 1 (N=298, 290) | 0.05 [0.05 to 0.05] | 0.05 [0.05 to 0.05]
  Day 8 (N= 297, 290) | 0.23 [0.21 to 0.25] | 0.13 [0.12 to 0.14]
  Day 15 (N= 292, 289) | 19 [17 to 21] | 12 [11 to 13]
  Day 50 (N= 292, 281) | 5.04 [4.56 to 5.57] | 10 [9.48 to 12]
  Day 91 (N= 293, 290) | 2.54 [2.29 to 2.82] | 3.8 [3.42 to 4.21]
  Day 181 (N= 292, 289) | 1.73 [1.53 to 1.95] | 1.5 [1.32 to 1.69]
  Day 366 (N= 291, 283) | 1.73 [1.53 to 1.95] | 1.2 [1.06 to 1.36]

8. Secondary Outcome: Percentages of Subjects With Anti-RVNA Titer ≥0.5 IU/mL in Children and Adult Subjects, ≥ 1 Years of Age
Description: Immunogenicity was assessed in terms of the Percentages of Subjects With Anti-RVNA concentration ≥0.5 IU/mL at Days 8, 15, 50, 91, 181 and 366 in Children and Adult Subjects, ≥ 1 Years of Age
Time Frame: At Days 8, 15, 50, 91, 181 and 366
Population: Per Protocol Set (PPS): all subjects who correctly receive the vaccine doses, provided immunogenicity data at the relevant time points and were not excluded due to reasons defined prior to the analysis. This outcome measure is only applicable for the 4-sites, 1-week without HRIG and 2-sites, TRC without HRIG Groups.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 4-sites, 1-week Without HRIG | 2-sites, TRC Without HRIG
Number analyzed (Participants) | 298 | 290
Percentages of Subjects
  Day 8 (N= 297, 290) | 21 [16 to 26] | 10 [7 to 14]
  Day 15 (N= 292, 289) | 100 [99 to 100] | 100 [99 to 100]
  Day 50 (N= 292, 281) | 100 [99 to 100] | 100 [99 to 100]
  Day 91 (N= 293, 290) | 99 [97 to 100] | 100 [98 to 100]
  Day 181 (N= 292, 289) | 96 [93 to 98] | 96 [92 to 98]
  Day 366 (N= 291, 283) | 95 [92 to 97] | 87 [82 to 90]

9. Secondary Outcome: Number of Subjects Who Reported Solicited Local and Systemic Adverse Events After Any Vaccination
Description: Number of subjects Who Reported Solicited Local and Systemic Adverse Events After Any Vaccination
Time Frame: From day 1 to day 3; from day 4 to day 7; from day 8 to day 14; from day 29 to day 35(2-sites, TRC PEP, ID regimen)
Population: Solicited Safety Set- All subjects in the Exposed Population who provide post vaccination solicited adverse event data. The number of exposed set participants analyzed for safety is different from the Per Protocol Set (PPS) for immunogenicity.
Measure: Number; unit: Subjects
Arm/Group | 4-sites, 1-week WITHOUT HRIG | 4-sites, 1-week WITH HRIG | 2-sites, TRC WITHOUT HRIG | 2-sites, TRC WITH HRIG
Number analyzed (Participants) | 356 | 85 | 353 | 89
Subjects
  Injection site erythema(≥ 1 to ≤ 5 Y); Day 1 | 0 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  Injection site erythema(≥ 1 to ≤ 5 Y); Day 4 | 0 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  Injection site erythema(≥ 1 to ≤ 5 Y); Day 8 | 1 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  Injection site erythema(≥ 1 to ≤ 5 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 2 | NA — No data as only adults to be enrolled to this group
  Injection site induration(≥ 1 to ≤ 5 Y); Day 1 | 0 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  Injection site induration(≥ 1 to ≤ 5 Y); Day 4 | 0 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  Injection site induration(≥ 1 to ≤ 5 Y); Day 8 | 0 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  Injection site induration(≥ 1 to ≤ 5 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 1 | NA — No data as only adults to be enrolled to this group
  Injection site swelling (≥ 1 to ≤ 5 Y); Day 1 | 0 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  Injection site swelling (≥ 1 to ≤ 5 Y); Day 4 | 0 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  Injection site swelling (≥ 1 to ≤ 5 Y); Day 8 | 0 | NA — No data as only adults to be enrolled to this group | 2 | NA — No data as only adults to be enrolled to this group
  Injection site swelling (≥ 1 to ≤ 5 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 8 | NA — No data as only adults to be enrolled to this group
  Injection site erythema (≥ 6 to ≤ 17 Y); Day 1 | 0 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  Injection site erythema (≥ 6 to ≤ 17 Y); Day 4 | 0 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  Injection site erythema (≥ 6 to ≤ 17 Y); Day 8 | 1 | NA — No data as only adults to be enrolled to this group | 2 | NA — No data as only adults to be enrolled to this group
  Injection site erythema (≥ 6 to ≤ 17 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 8 | NA — No data as only adults to be enrolled to this group
  Injection site induration (≥ 6 to ≤ 17 Y); Day 1 | 0 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  Injection site induration (≥ 6 to ≤ 17 Y); Day 4 | 1 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  Injection site induration (≥ 6 to ≤ 17 Y); Day 8 | 0 | NA — No data as only adults to be enrolled to this group | 1 | NA — No data as only adults to be enrolled to this group
  Injection site induration (≥ 6 to ≤ 17 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 2 | NA — No data as only adults to be enrolled to this group
  Injection site swelling (≥ 6 to ≤ 17 Y); Day 1 | 0 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  Injection site swelling (≥ 6 to ≤ 17 Y); Day 4 | 1 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  Injection site swelling (≥ 6 to ≤ 17 Y); Day 8 | 0 | NA — No data as only adults to be enrolled to this group | 2 | NA — No data as only adults to be enrolled to this group
  Injection site swelling (≥ 6 to ≤ 17 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 2 | NA — No data as only adults to be enrolled to this group
  Injection site erythema (≥ 18 Y); Day 1 | 3 | 6 | 2 | 3
  Injection site erythema (≥ 18 Y); Day 4 | 11 | 4 | 4 | 5
  Injection site erythema (≥ 18 Y); Day 8 | 12 | 1 | 8 | 4
  Injection site erythema (≥ 18 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — Not assessed at Day 29 for this group | 27 | 13
  Injection site induration (≥ 18 Y); Day 1 | 0 | 0 | 0 | 0
  Injection site induration (≥ 18 Y); Day 4 | 0 | 0 | 0 | 0
  Injection site induration (≥ 18 Y); Day 8 | 2 | 0 | 2 | 0
  Injection site induration (≥ 18 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — Not assessed at Day 29 for this group | 4 | 1
  Injection site swelling (≥ 18 Y); Day 1 | 0 | 0 | 1 | 0
  Injection site swelling (≥ 18 Y); Day 4 | 0 | 0 | 0 | 0
  Injection site swelling (≥ 18 Y); Day 8 | 0 | 0 | 2 | 0
  Injection site swelling (≥ 18 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — Not assessed at Day 29 for this group | 5 | 1
  Change In Eating Habits,( ≥ 1 to ≤ 5 Y); Day 1 | 4 | NA — No data as only adults to be enrolled to this group | 3 | NA — No data as only adults to be enrolled to this group
  Change In Eating Habits,( ≥ 1 to ≤ 5 Y); Day 4 | 3 | NA — No data as only adults to be enrolled to this group | 1 | NA — No data as only adults to be enrolled to this group
  Change In Eating Habits,( ≥ 1 to ≤ 5 Y); Day 8 | 3 | NA — No data as only adults to be enrolled to this group | 2 | NA — No data as only adults to be enrolled to this group
  Change In Eating Habits,( ≥ 1 to ≤ 5 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 6 | NA — No data as only adults to be enrolled to this group
  Sleepiness (≥ 1 to ≤ 5 Y); Day 1 | 4 | NA — No data as only adults to be enrolled to this group | 7 | NA — No data as only adults to be enrolled to this group
  Sleepiness (≥ 1 to ≤ 5 Y); Day 4 | 7 | NA — No data as only adults to be enrolled to this group | 3 | NA — No data as only adults to be enrolled to this group
  Sleepiness (≥ 1 to ≤ 5 Y); Day 8 | 2 | NA — No data as only adults to be enrolled to this group | 4 | NA — No data as only adults to be enrolled to this group
  Sleepiness (≥ 1 to ≤ 5 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 2 | NA — No data as only adults to be enrolled to this group
  Vomiting (≥ 1 to ≤ 5 Y); Day 1 | 4 | NA — No data as only adults to be enrolled to this group | 1 | NA — No data as only adults to be enrolled to this group
  Vomiting (≥ 1 to ≤ 5 Y); Day 4 | 2 | NA — No data as only adults to be enrolled to this group | 1 | NA — No data as only adults to be enrolled to this group
  Vomiting (≥ 1 to ≤ 5 Y); Day 8 | 1 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  Vomiting (≥ 1 to ≤ 5 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 5 | NA — No data as only adults to be enrolled to this group
  Diarrhea (≥ 1 to ≤ 5 Y); Day 1 | 3 | NA — No data as only adults to be enrolled to this group | 2 | NA — No data as only adults to be enrolled to this group
  Diarrhea (≥ 1 to ≤ 5 Y); Day 4 | 2 | NA — No data as only adults to be enrolled to this group | 2 | NA — No data as only adults to be enrolled to this group
  Diarrhea (≥ 1 to ≤ 5 Y); Day 8 | 4 | NA — No data as only adults to be enrolled to this group | 1 | NA — No data as only adults to be enrolled to this group
  Diarrhea (≥ 1 to ≤ 5 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 4 | NA — No data as only adults to be enrolled to this group
  Irritability.( ≥ 1 to ≤ 5 Y); Day 1 | 5 | NA — No data as only adults to be enrolled to this group | 3 | NA — No data as only adults to be enrolled to this group
  Irritability.( ≥ 1 to ≤ 5 Y); Day 4 | 3 | NA — No data as only adults to be enrolled to this group | 3 | NA — No data as only adults to be enrolled to this group
  Irritability.( ≥ 1 to ≤ 5 Y); Day 8 | 1 | NA — No data as only adults to be enrolled to this group | 5 | NA — No data as only adults to be enrolled to this group
  Irritability.( ≥ 1 to ≤ 5 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 5 | NA — No data as only adults to be enrolled to this group
  Chills(≥ 6 to ≤ 17 Y); Day 1 | 2 | NA — No data as only adults to be enrolled to this group | 2 | NA — No data as only adults to be enrolled to this group
  Chills(≥ 6 to ≤ 17 Y); Day 4 | 0 | NA — No data as only adults to be enrolled to this group | 1 | NA — No data as only adults to be enrolled to this group
  Chills(≥ 6 to ≤ 17 Y); Day 8 | 1 | NA — No data as only adults to be enrolled to this group | 1 | NA — No data as only adults to be enrolled to this group
  Chills(≥ 6 to ≤ 17 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  Nausea ( ≥ 6 to ≤ 17 Y); Day 1 | 4 | NA — No data as only adults to be enrolled to this group | 3 | NA — No data as only adults to be enrolled to this group
  Nausea ( ≥ 6 to ≤ 17 Y); Day 4 | 2 | NA — No data as only adults to be enrolled to this group | 1 | NA — No data as only adults to be enrolled to this group
  Nausea ( ≥ 6 to ≤ 17 Y); Day 8 | 3 | NA — No data as only adults to be enrolled to this group | 1 | NA — No data as only adults to be enrolled to this group
  Nausea ( ≥ 6 to ≤ 17 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  Generalized Myalgia (≥ 6 to ≤ 17 Y); Day 1 | 5 | NA — No data as only adults to be enrolled to this group | 1 | NA — No data as only adults to be enrolled to this group
  Generalized Myalgia (≥ 6 to ≤ 17 Y); Day 4 | 4 | NA — No data as only adults to be enrolled to this group | 2 | NA — No data as only adults to be enrolled to this group
  Generalized Myalgia (≥ 6 to ≤ 17 Y); Day 8 | 2 | NA — No data as only adults to be enrolled to this group | 3 | NA — No data as only adults to be enrolled to this group
  Generalized Myalgia (≥ 6 to ≤ 17 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 4 | NA — No data as only adults to be enrolled to this group
  Generalized Arthralgia (≥ 6 to ≤ 17 Y); Day 1 | 3 | NA — No data as only adults to be enrolled to this group | 1 | NA — No data as only adults to be enrolled to this group
  Generalized Arthralgia (≥ 6 to ≤ 17 Y); Day 4 | 1 | NA — No data as only adults to be enrolled to this group | 1 | NA — No data as only adults to be enrolled to this group
  Generalized Arthralgia (≥ 6 to ≤ 17 Y); Day 8 | 4 | NA — No data as only adults to be enrolled to this group | 2 | NA — No data as only adults to be enrolled to this group
  Generalized Arthralgia (≥ 6 to ≤ 17 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 1 | NA — No data as only adults to be enrolled to this group
  Headache (≥ 6 to ≤ 17 Y); Day 1 | 8 | NA — No data as only adults to be enrolled to this group | 9 | NA — No data as only adults to be enrolled to this group
  Headache (≥ 6 to ≤ 17 Y); Day 4 | 8 | NA — No data as only adults to be enrolled to this group | 8 | NA — No data as only adults to be enrolled to this group
  Headache (≥ 6 to ≤ 17 Y); Day 8 | 6 | NA — No data as only adults to be enrolled to this group | 6 | NA — No data as only adults to be enrolled to this group
  Headache (≥ 6 to ≤ 17 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 3 | NA — No data as only adults to be enrolled to this group
  Fatigue (≥ 6 to ≤ 17 Y); Day 1 | 8 | NA — No data as only adults to be enrolled to this group | 7 | NA — No data as only adults to be enrolled to this group
  Fatigue (≥ 6 to ≤ 17 Y); Day 4 | 5 | NA — No data as only adults to be enrolled to this group | 1 | NA — No data as only adults to be enrolled to this group
  Fatigue (≥ 6 to ≤ 17 Y); Day 8 | 1 | NA — No data as only adults to be enrolled to this group | 6 | NA — No data as only adults to be enrolled to this group
  Fatigue (≥ 6 to ≤ 17 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 6 | NA — No data as only adults to be enrolled to this group
  Rash (≥ 6 to ≤ 17 Y); Day 1 | 4 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  Rash (≥ 6 to ≤ 17 Y); Day 4 | 3 | NA — No data as only adults to be enrolled to this group | 3 | NA — No data as only adults to be enrolled to this group
  Rash (≥ 6 to ≤ 17 Y); Day 8 | 3 | NA — No data as only adults to be enrolled to this group | 3 | NA — No data as only adults to be enrolled to this group
  Rash (≥ 6 to ≤ 17 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 2 | NA — No data as only adults to be enrolled to this group
  Vomitting (≥ 6 to ≤ 17 Y); Day 1 | 3 | NA — No data as only adults to be enrolled to this group | 5 | NA — No data as only adults to be enrolled to this group
  Vomitting (≥ 6 to ≤ 17 Y); Day 4 | 2 | NA — No data as only adults to be enrolled to this group | 1 | NA — No data as only adults to be enrolled to this group
  Vomitting (≥ 6 to ≤ 17 Y); Day 8 | 3 | NA — No data as only adults to be enrolled to this group | 2 | NA — No data as only adults to be enrolled to this group
  Vomitting (≥ 6 to ≤ 17 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 1 | NA — No data as only adults to be enrolled to this group
  Diarrhea (≥ 6 to ≤ 17 Y); Day 1 | 4 | NA — No data as only adults to be enrolled to this group | 2 | NA — No data as only adults to be enrolled to this group
  Diarrhea (≥ 6 to ≤ 17 Y); Day 4 | 0 | NA — No data as only adults to be enrolled to this group | 1 | NA — No data as only adults to be enrolled to this group
  Diarrhea (≥ 6 to ≤ 17 Y); Day 8 | 1 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  Diarrhea (≥ 6 to ≤ 17 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  Loss Of Appetite (≥ 6 to ≤ 17 Y); Day 1 | 6 | NA — No data as only adults to be enrolled to this group | 3 | NA — No data as only adults to be enrolled to this group
  Loss Of Appetite (≥ 6 to ≤ 17 Y); Day 4 | 3 | NA — No data as only adults to be enrolled to this group | 1 | NA — No data as only adults to be enrolled to this group
  Loss Of Appetite (≥ 6 to ≤ 17 Y); Day 8 | 1 | NA — No data as only adults to be enrolled to this group | 1 | NA — No data as only adults to be enrolled to this group
  Loss Of Appetite (≥ 6 to ≤ 17 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  Chills (≥ 18 Y); Day 1 | 8 | 3 | 5 | 2
  Chills (≥ 18 Y); Day 4 | 1 | 2 | 6 | 4
  Chills (≥ 18 Y); Day 8 | 5 | 0 | 4 | 0
  Chills (≥ 18 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — Not assessed at Day 29 for this group | 0 | 0
  Nausea,( ≥ 18 Y); Day 1 | 8 | 3 | 3 | 3
  Nausea,( ≥ 18 Y); Day 4 | 4 | 2 | 2 | 3
  Nausea,( ≥ 18 Y); Day 8 | 4 | 0 | 4 | 3
  Nausea,( ≥ 18 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — Not assessed at Day 29 for this group | 0 | 0
  Generalized Myalgia (≥ 18 Y); Day 1 | 23 | 12 | 19 | 12
  Generalized Myalgia (≥ 18 Y); Day 4 | 16 | 7 | 12 | 6
  Generalized Myalgia (≥ 18 Y); Day 8 | 20 | 5 | 15 | 9
  Generalized Myalgia (≥ 18 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — Not assessed at Day 29 for this group | 7 | 4
  Generalized Arthralgia (≥ 18 Y); Day 1 | 18 | 7 | 13 | 7
  Generalized Arthralgia (≥ 18 Y); Day 4 | 6 | 5 | 10 | 7
  Generalized Arthralgia (≥ 18 Y); Day 8 | 15 | 3 | 15 | 6
  Generalized Arthralgia (≥ 18 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — Not assessed at Day 29 for this group | 6 | 4
  Headache (≥ 18 Y); Day 1 | 24 | 6 | 11 | 13
  Headache (≥ 18 Y); Day 4 | 14 | 10 | 15 | 11
  Headache (≥ 18 Y); Day 8 | 19 | 8 | 15 | 16
  Headache (≥ 18 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — Not assessed at Day 29 for this group | 12 | 11
  Fatigue (≥ 18 Y); Day 1 | 28 | 11 | 19 | 10
  Fatigue (≥ 18 Y); Day 4 | 21 | 6 | 17 | 11
  Fatigue (≥ 18 Y); Day 8 | 19 | 8 | 15 | 14
  Fatigue (≥ 18 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — Not assessed at Day 29 for this group | 9 | 10
  Rash (≥ 18 Y); Day 1 | 10 | 3 | 4 | 0
  Rash (≥ 18 Y); Day 4 | 4 | 3 | 8 | 4
  Rash (≥ 18 Y); Day 8 | 6 | 4 | 11 | 2
  Rash (≥ 18 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — Not assessed at Day 29 for this group | 2 | 2
  Vomitting (≥ 18 Y); Day 1 | 0 | 0 | 2 | 0
  Vomitting (≥ 18 Y); Day 4 | 0 | 1 | 1 | 1
  Vomitting (≥ 18 Y); Day 8 | 1 | 0 | 1 | 3
  Vomitting (≥ 18 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — Not assessed at Day 29 for this group | 1 | 0
  Diarrhea (≥ 18 Y); Day 1 | 5 | 4 | 2 | 5
  Diarrhea (≥ 18 Y); Day 4 | 3 | 2 | 5 | 3
  Diarrhea (≥ 18 Y); Day 8 | 5 | 1 | 4 | 4
  Diarrhea (≥ 18 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — Not assessed at Day 29 for this group | 3 | 0
  Loss Of Appetite (≥ 18 Y); Day 1 | 7 | 0 | 5 | 2
  Loss Of Appetite (≥ 18 Y); Day 4 | 3 | 2 | 2 | 0
  Loss Of Appetite (≥ 18 Y); Day 8 | 3 | 3 | 2 | 4
  Loss Of Appetite (≥ 18 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — Not assessed at Day 29 for this group | 1 | 1
  Injection site tenderness (≥ 1 to ≤ 5 Y); Day 1 | 15 | NA — No data as only adults to be enrolled to this group | 8 | NA — No data as only adults to be enrolled to this group
  Injection site tenderness (≥ 1 to ≤ 5 Y); Day 4 | 8 | NA — No data as only adults to be enrolled to this group | 9 | NA — No data as only adults to be enrolled to this group
  Injection site tenderness (≥ 1 to ≤ 5 Y); Day 8 | 7 | NA — No data as only adults to be enrolled to this group | 8 | NA — No data as only adults to be enrolled to this group
  Injection site tenderness (≥ 1 to ≤ 5 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 9 | NA — No data as only adults to be enrolled to this group
  Injection site pain (≥ 6 to ≤ 17 Y); Day 1 | 14 | NA — No data as only adults to be enrolled to this group | 7 | NA — No data as only adults to be enrolled to this group
  Injection site pain (≥ 6 to ≤ 17 Y); Day 4 | 6 | NA — No data as only adults to be enrolled to this group | 10 | NA — No data as only adults to be enrolled to this group
  Injection site pain (≥ 6 to ≤ 17 Y); Day 8 | 6 | NA — No data as only adults to be enrolled to this group | 11 | NA — No data as only adults to be enrolled to this group
  Injection site pain (≥ 6 to ≤ 17 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — No data as only adults to be enrolled to this group | 6 | NA — No data as only adults to be enrolled to this group
  Injection site pain (≥ 18 Y); Day 1 | 12 | 6 | 16 | 11
  Injection site pain (≥ 18 Y); Day 4 | 8 | 8 | 13 | 3
  Injection site pain (≥ 18 Y); Day 8 | 8 | 7 | 21 | 3
  Injection site pain (≥ 18 Y); Day 29 | NA — Not assessed at Day 29 for this group | NA — Not assessed at Day 29 for this group | 14 | 9

10. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: Safety was assessed in terms of the Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Time Frame: Day 1 to Day 366
Population: Unsolicited Safety Set- All subjects in the Exposed Population who have post vaccination unsolicited adverse event records. The number of exposed set participants analyzed for safety is different from the Per Protocol Set (PPS) for immunogenicity.
Measure: Number; unit: Subjects
Arm/Group | 4-sites, 1-week WITHOUT HRIG | 4-sites, 1-week WITH HRIG | 2-sites, TRC WITHOUT HRIG | 2-sites, TRC WITH HRIG
Number analyzed (Participants) | 356 | 85 | 353 | 89
Subjects
  ≥ 1 to ≤ 5 Y Any AEs;D1-366 | 45 | NA — No data as only adults to be enrolled to this group | 53 | NA — No data as only adults to be enrolled to this group
  ≥ 1 to ≤ 5 Y SAE;D1-366 | 3 | NA — No data as only adults to be enrolled to this group | 4 | NA — No data as only adults to be enrolled to this group
  ≥ 1 to ≤ 5 Y At least possibly related SAEs;D1-366 | 0 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  ≥ 1 to ≤ 5 Y Deaths;D1-366 | 0 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  ≥1 to ≤ 5 Y Withdrawal from study due to AE;D1-366 | 0 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  ≥ 6 to ≤ 17 Y Any AEs;D1-366 | 58 | NA — No data as only adults to be enrolled to this group | 71 | 1
  ≥ 6 to ≤ 17 Y SAE;D1-366 | 1 | NA — No data as only adults to be enrolled to this group | 3 | NA — No data as only adults to be enrolled to this group
  ≥6 to ≤ 17 Y At least possibly related SAEs;D1-366 | 0 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  ≥ 6 to ≤ 17 Y Deaths;D1-366 | 0 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  ≥6 to ≤17 Y Withdrawal from study due to AE;D1-366 | 0 | NA — No data as only adults to be enrolled to this group | 0 | NA — No data as only adults to be enrolled to this group
  ≥ 18 Y Any AEs;D1-366 | 157 | 71 | 156 | 72
  ≥ 18 Y SAE;D1-366 | 8 | 3 | 7 | 5
  ≥ 18 Y At least possibly related SAEs;D1-366 | 0 | 0 | 0 | 0
  ≥ 18 Y Deaths;D1-366 | 0 | 0 | 0 | 0
  ≥ 18 Y Withdrawal from study due to AE;D1-366 | 0 | 0 | 0 | 0
  Overall population ≥ 1 Y Any AEs;D1-366 | 260 | 71 | 280 | 73
  Overall population ≥ 1 Y SAE;D1-366 | 12 | 3 | 14 | 5
  Overall ≥1Y Atleast possibly related SAEs;D1-366 | 0 | 0 | 0 | 0
  Overall population ≥ 1 Y Deaths;D1-366 | 0 | 0 | 0 | 0
  Overall population ≥1Y Withdrawal due to AE;D1-366 | 0 | 0 | 0 | 0

11. Secondary Outcome: Geometric Mean Rabies Virus Neutralizing Antibody (RVNA) Concentration ≥0.5 IU/mL and Vaccine Group Differences in Adult Subjects, ≥ 18 Years of Age
Description: Immunogenicity was assessed in terms of the Geometric Mean Rabies Virus Neutralizing Antibody (RVNA) Concentration ≥0.5 IU/mL at Days 8, 15, 50,91, 181 and 366 in Adult Subjects, ≥ 18 Years of Age
Time Frame: At Days 8, 15, 50, 91, 181 and 366
Population: Per Protocol Set (PPS): all subjects who correctly receive the vaccine doses, provided immunogenicity data at the relevant time points and were not excluded due to reasons defined prior to the analysis. This outcome measure is applicable only for 4-sites, 1-week with HRIG and 2-sites TRC with HRIG Groups.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Groups:
- 2-sites TRC WITH HRIG: 8 doses of the PCEC rabies vaccine, administered ID (0.1ml for each injection) to adults only, according to the "2-sites, TRC", updated Thai Red Cross regimen, with or without HRIG administered on day 1
Arm/Group | 4-sites, 1-week WITH HRIG | 2-sites TRC WITH HRIG
Number analyzed (Participants) | 66 | 72
IU/mL
  Day 1 (N= 66, 72) | 0.05 [0.05 to 0.05] | 0.05 [0.05 to 0.05]
  Day 8 (N= 66, 72) | 0.21 [0.17 to 0.26] | 0.17 [0.14 to 0.21]
  Day 15 (N= 65, 72) | 13 [11 to 15] | 8.37 [6.96 to 10]
  Day 50 (N= 65, 69) | 1.97 [1.6 to 2.43] | 6.37 [5.21 to 7.78]
  Day 91 (N= 65, 72) | 1.01 [0.81 to 1.27] | 2.25 [1.81 to 2.79]
  Day 181 (N= 65, 71) | 0.88 [0.67 to 1.14] | 1.05 [0.81 to 1.35]
  Day 366 (N= 65, 69) | 0.68 [0.53 to 0.88] | 0.59 [0.46 to 0.76]

12. Secondary Outcome: Percentages of Subjects With Anti-RVNA Titer ≥0.5 IU/mL in Adult Subjects, ≥ 18 Years of Age
Description: Immunogenicity was assessed in terms of the number of subjects With Anti-RVNA concentration ≥0.5 IU/mL at Days 8, 15, 50, 91, 181 and 366 in Adult Subjects, ≥ 18 Years of Age
Time Frame: At Days 8, 15,50, 91, 181 and 366
Population: Per Protocol Set (PPS): all subjects who correctly receive the vaccine doses, provided immunogenicity data at the relevant time points and were not excluded due to reasons defined prior to the analysis. This outcome measure is applicable only for 4-sites, 1-week with HRIG and 2-sites, TRC with HRIG Groups
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Groups:
- 2-sites, TRC WITH HRIG: 8 doses of the PCEC rabies vaccine, administered ID (0.1ml for each injection) to adults only, according to the "2-sites, TRC", updated Thai Red Cross regimen, with or without HRIG administered on day 1
Arm/Group | 4-sites, 1-week WITH HRIG | 2-sites, TRC WITH HRIG
Number analyzed (Participants) | 66 | 72
Percentages of Subjects
  Day 1 (N= 66, 72) | 0 [0 to 5] | 0 [0 to 5]
  Day 8 (N= 66, 72) | 8 [3 to 17] | 10 [4 to 19]
  Day 15 (N= 65, 72) | 100 [94 to 100] | 99 [93 to 100]
  Day 50 (N= 65, 69) | 95 [87 to 99] | 100 [95 to 100]
  Day 91 (N= 65, 72) | 83 [72 to 91] | 99 [93 to 100]
  Day 181 (N= 65, 71) | 77 [65 to 86] | 85 [74 to 92]
  Day 366 (N= 65, 69) | 66 [53 to 77] | 70 [57 to 80]

ADVERSE EVENTS:
Time Frame: Day 1 to day 366 (Study Groups: A1- 4-sites, 1-week" (4-4-4-0-0) ID PEP regimen without HRIG, A2- 4-sites, 1-week" (4-4-4-0-0) ID PEP regimen with HRIG, B1- 2-sites TRC" (2-2-2-0-2) ID PEP regimen without HRIG, B2- 2-sites TRC" (2-2-2-0-2) ID PEP regimen with HRIG).
Description: Solicited local,systemic AEs & associated medications will be recorded on diary cards for 3,4, 7 & 7 days post vaccination on Visits 1,2,3 & 5,respectively.Unsolicited AEs & associated vaccinations will be collected in diary cards from D1-29 for Groups A1 & A2 & from D1-50 for Groups B1 & B2.After D29/50, until D366 only SAEs & AEs leading to withdrawal & associated vaccinations will be recorded.Number of exposed set participants analyzed for safety is different from the PPS for immunogenicity.
Arm/Group | 4-sites, 1-week WITHOUT HRIG | 4-sites, 1-week WITH HRIG | 2-sites, TRC WITHOUT HRIG | 2-sites, TRC WITH HRIG
Serious Adverse Events (participants affected / at risk) | 5/356 | 1/85 | 4/353 | 2/89
Other Adverse Events (participants affected / at risk) | 292/356 | 78/85 | 298/353 | 82/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 4-sites, 1-week WITHOUT HRIG (N=356) | 4-sites, 1-week WITH HRIG (N=85) | 2-sites, TRC WITHOUT HRIG (N=353) | 2-sites, TRC WITH HRIG (N=89)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Angina Unstable (Cardiac disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Irritable Bowel Syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Appendiceal Abscess (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis Perforated (Infections and infestations) | 1 | 0 | 0 | 0
Dengue Fever (Infections and infestations) | 1 | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
HIV Infection (Infections and infestations) | 1 | 0 | 0 | 0
Hand-Foot-And-Mouth Disease (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Immune system disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pseudomonal Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Animal Bite (Injury, poisoning and procedural complications) | 5 | 0 | 4 | 2
Animal Scratch (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Dysfunctional Uterine Bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 4-sites, 1-week WITHOUT HRIG (N=356) | 4-sites, 1-week WITH HRIG (N=85) | 2-sites, TRC WITHOUT HRIG (N=353) | 2-sites, TRC WITH HRIG (N=89)
DIARRHOEA (Gastrointestinal disorders) | 28 | 8 | 20 | 8
NAUSEA (Gastrointestinal disorders) | 22 | 4 | 12 | 7
VOMITING (Gastrointestinal disorders) | 15 | 1 | 20 | 4
CHILLS (General disorders) | 15 | 4 | 13 | 5
FATIGUE (General disorders) | 53 | 16 | 52 | 24
INJECTION SITE ERYTHEMA (General disorders) | 195 | 59 | 168 | 56
INJECTION SITE INDURATION (General disorders) | 52 | 13 | 62 | 13
INJECTION SITE PAIN (General disorders) | 77 | 18 | 89 | 20
INJECTION SITE SWELLING (General disorders) | 39 | 8 | 47 | 4
PYREXIA (General disorders) | 15 | 3 | 27 | 4
VACCINATION SITE ERYTHEMA (General disorders) | 82 | 19 | 79 | 23
VACCINATION SITE INDURATION (General disorders) | 26 | 5 | 22 | 7
VACCINATION SITE SWELLING (General disorders) | 13 | 5 | 19 | 2
NASOPHARYNGITIS (Infections and infestations) | 13 | 1 | 28 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 19 | 6 | 28 | 5
DECREASED APPETITE (Metabolism and nutrition disorders) | 19 | 5 | 12 | 7
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 33 | 9 | 33 | 17
MYALGIA (Musculoskeletal and connective tissue disorders) | 45 | 19 | 41 | 19
HEADACHE (Nervous system disorders) | 53 | 21 | 54 | 31
RASH (Skin and subcutaneous tissue disorders) | 21 | 7 | 24 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreement with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publications of the pooled data (i.e., data from all sites) in the clinical trial.